CLINICAL TRIAL: NCT05151107
Title: Relationship Between Residual Gastric Area and Weight Loss After Sleeve Gastrectomy: a Cohort Study
Brief Title: Residual Gastric Area and Weight Loss After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical doctor, University of Foggia
Other Study IDs: 1
Record Dates: First submitted 2021-11-15; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The radiographic images were collected through a software called "PACS" which combined with a viewer for image processing, that allows the calculation of the residual stomach area (RSA). — Upper gastrointestinal radiographie

SUMMARY:
BACKGROUND: The aim of this study is to evaluate the impact of the actual size and area of the remnant stomach, as measured by Upper gastrointestinal tract radiography, on weight loss after LSG.

MATERIALS AND METHODS: From May 2017 to December 2019, 56 patients with morbid obesity were admitted to the Department of Medical and Surgical Sciences, University of Foggia and underwent laparoscopic sleeve gastrectomy.

UGI tract radiography was performed on day two after the operation to rule out leakage.

DETAILED DESCRIPTION:
Study design and setting

From May 2017 to December 2019, 56 patients with morbid obesity were admitted to the Department of Medical and Surgical Sciences, University of Foggia and underwent laparoscopic sleeve gastrectomy. UGI tract radiography with water-soluble contrast medium was performed on the second day after the operation to rule out leakage. The radiographic images were collected through a software program called "PACS" which combined with a viewer for image processing, allows for the calculation of the residual stomach area (RSA). RSA was correlated with postoperative weight (EWL) at 1, 6, and 12 months.

Eligibility criteria

Adult patients of both genders with morbid obesity defined as BMI>40 kg/m2 or BMI>35 kg/m2 with at least one associated major comorbidity were included. We excluded patients with secondary obesity due to endocrine and psychological disorders, patients with previous bariatric procedures and patients unwilling to comply with postoperative diet and exercise program.

Statistical analysis

Continuous data were expressed as mean and standard deviation (SD) and they were analyzed using Student's T test. The correlation between gastric volume before and after LSG and BMI and weight loss was measured using Pearson correlation coefficient test. Correlation coefficients were classified as strong (-1.0 to -0.5 or 0.5 to 1.0), moderate (-0.5 to -0.3 or 0.3 to 0.5), and weak (-0.3 to -0.1 or 0.1 to 0.3). P<0.05 was considered statistically significant. This work is fully compliant with the STROCSS criteria

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders with morbid obesity defined as BMI>40 kg/m2
* Adult patients of both genders with morbid obesity defined as BMI>35 kg/m2 with at least one associated major comorbidity

Exclusion Criteria:

* Patients with secondary obesity due to endocrine and psychologic disorders
* Patients whit previous bariatric procedures
* Patients unwilling to comply with postoperative diet regimen and exercise program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 56 patients underwent sleeve gastrectomy with a mean age of 43,5± 11 years of which 40 were female.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Postoperative EWL % correlated with the Residual Stomach Area | 2017-2019
  the impact of the actual size and area of the remnant stomach, as measured by Upper gastrointestinal tract radiography, on weight loss

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Giovanna Pavone, Foggia
  - Nicola Tartaglia, Foggia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT05151107/Prot_SAP_000.pdf